CLINICAL TRIAL: NCT00305851
Title: Stories and Music for Adolescent/Young Adult Resilience During Transplant (SMART)
Brief Title: Music Therapy or Book Discussion in Improving Quality of Life in Young Patients Undergoing Stem Cell Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COG-ANUR0631; NCI-2009-00408 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000463879; COG-ANUR0631 (Other: Children's Oncology Group); COG-ANUR0631 (Other: DCP); ANUR0631 (Other: CTEP); R01NR008583 (NIH); U10CA095861 (NIH)
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2022-07-15 (Actual); Status verified 2013-01

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Music Therapy; Psychiatric Rehabilitation

ARMS (2):
- Arm I (counseling) (Active Comparator): Patients undergo six 1-hour sessions twice a week for 3 weeks with a trained counselor in which they choose up to 3 books on CD and listen to the book and/or discuss their impressions and thoughts about the contents with the counselor. Patients are provided with a portable CD player to listen to the books during their hospitalization.
  Interventions: Procedure: Psychosocial Assessment and Care; Other: Quality-of-Life Assessment
- Arm II (counseling and music therapy) (Experimental): Patients undergo six 1-hour sessions twice a week for 3 weeks with a music therapist, designed specifically for the pre-transplant and acute phase of treatment. Phases of patient participation include song writing, recording the song with a digital accompaniment track, completing a video layout worksheet, taking photos or making drawings for the video, viewing clip art and pictures on a computer, and sharing the final video with family members and hospital staff.
  Interventions: Procedure: Music Therapy; Procedure: Psychosocial Assessment and Care; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Music Therapy — Undergo therapeutic music video therapy
  Arms: Arm II (counseling and music therapy)
Procedure: Psychosocial Assessment and Care — Undergo books on tape therapy
  Other Names: Psychosocial Care/Assessment
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial is studying how well music therapy works compared to listening and discussing books on tape in improving quality of life in young patients undergoing stem cell transplant. Music therapy or book discussion may improve quality of life in patients undergoing stem cell transplant. It is not yet known whether music therapy is more effective than book discussion in improving quality of life in patients undergoing stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test the efficacy, in terms of resilience and quality of life, of a therapeutic music video (TMV) intervention vs listening and discussing books on tape (control group) for adolescents and young adults (AYA) undergoing autologous or allogeneic transplantation for cancer.

II. Qualitatively describe the perception of helpfulness and meaningfulness of a sub-group of both interventions for AYA and family members 100 days post-transplant.

OUTLINE: This is a randomized, controlled, limited multicenter study. Patients are randomized to 1 of 2 arms.

ARM I (books on tape [control group]): Patients undergo six 1-hour sessions twice a week for 3 weeks with a trained counselor in which they choose up to 3 books on CD and listen to the book and/or discuss their impressions and thoughts about the contents with the counselor. Patients are provided with a portable CD player to listen to the books during their hospitalization.

ARM II (therapeutic music video [TMV] intervention): Patients undergo six 1-hour sessions twice a week for 3 weeks with a music therapist, designed specifically for the pre-transplant and acute phase of treatment. Phases of patient participation include song writing, recording the song with a digital accompaniment track, completing a video layout worksheet, taking photos or making drawings for the video, viewing clip art and pictures on a computer, and sharing the final video with family members and hospital staff.

In both arms, patients complete questionnaires before and after sessions 2, 4, and 6 with the music therapist. Patients also complete computer-based questionnaires before hospitalization, after session six during hospitalization, and at 100 days post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an oncology condition requiring allogeneic or autologous transplantation
* Receiving or planning to receive a myeloablative treatment regimen and 1 of the following:

  * Marrow transplantation
  * Peripheral stem cell transplantation
  * Cord blood stem cell transplantation
* Patients with cancers that do not usually occur in childhood/adolescent or young adult populations (e.g., breast or prostate cancer) are not eligible
* Able to read and speak English

  * English does not need to be the primary language
* Able to participate in the sessions as evaluated for alertness and engagement by the music therapist
* No cognitive impairments that would make it difficult to participate in the intervention or complete questionnaires
* Not married and not a parent
* Concurrent therapy for pain control or relief of other symptoms allowed

Ages: 11 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 118 (Actual)
Dates: Start 2006-04-15 (Actual); Primary Completion 2010-10-05 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Assess acute changes of Symptoms-related distress: Pain | Change from pre- and post-sessions 2, 4, and 6, baseline, immediately after completion of study treatment, and 100 days post-transplant
  Illness-related distress will be measured by indicators of uncertainty in illness, symptom-related distress. Brief Symptoms Assessment is a self-reported measure capturing information on pain. Specifically, the instrument includes a 1-item pain numeric rating scale.
Assess acute changes of Symptoms-related distress: Anxiety | Change from pre- and post-sessions 2, 4, and 6, baseline, immediately after completion of study treatment, and 100 days post-transplant
  Illness-related distress will be measured by indicators of uncertainty in illness, symptom-related distress. Brief Symptoms Assessment is a self-reported measure capturing information on anxiety. Specifically, the instrument includes a 5-item Anxiety scale.
Assess acute changes of Symptoms-related distress: Fatigue | Change from pre- and post-sessions 2, 4, and 6, baseline, immediately after completion of study treatment, and 100 days post-transplant
  Illness-related distress will be measured by indicators of uncertainty in illness, symptom-related distress. Brief Symptoms Assessment is a self-reported measure capturing information on fatigue. Specifically, the instrument includes a 1-item fatigue visual analogue scale.
Assess acute changes of Symptoms-related distress: Mood | Change from pre- and post-sessions 2, 4, and 6, baseline, immediately after completion of study treatment, and 100 days post-transplant
  Illness-related distress will be measured by indicators of uncertainty in illness, symptom-related distress. Brief Symptoms Assessment is a self-reported measures capturing information on mood. Specifically, the instrument includes a 1-item mood scale.
Assess changes in uncertainty in illness as assessed by the Mishel Uncertainty in Illness Scale | Change from baseline, immediately after completion of study treatment and 100 days post-transplant
  Mishel Uncertainty in Illness Scale-Revised (MUIS-R) consists of two factors: Complexity and Ambiguity, with higher scores indicating a high level of uncertainty. Item responses are on a 5-point Likert-type scale (ranging from 5 = Strongly Agree to 1 = Strongly Disagree
Assess changes in the use of defensive coping | Change from immediately after completion of study treatment and 100 days post-transplant
  Defensive Coping will be measured by three subscales of the Jalowiec Coping Scale-Revised (JCS):
  evasive, emotive, and fatalistic coping. JCS is a self-report, 0-3 point rating scale. The items are scored for both use and effectiveness.
Assess changes in the use of positive coping | Change from immediately after completion of study treatment and 100 days post-transplant
  Three subscales of the Jalowiec Coping Scale-Revised will measure Positive Coping (JCS): confrontive, optimistic, and supportive.
Assess changes in communication with family as assessed by Parent-Adolescent Communication | Change from baseline, immediately after completion of study treatment, and 100 days post-transplant
  Parent Adolescent Communication (P-AC) self-report items are on 5-point Likert scales that assess adolescents' views regarding their perceptions and experience of communicating with each parent rated separately. The two subscales, Open Family Communication and Problems in Family Communication, respectively measure positive and negative aspects of communications within a family and are scored independently.
Assess changes in adaptability or cohesion as assessed by FACES II | Change from baseline, immediately after completion of study treatment, and 100 days post-transplant
  Family Adaptability and Cohesion Scale II (FACES II) is a self-report scale using Likert response scales and measuring the 2 factors: Adaptability or cohesion
Assess changes in perceived social support from friends | Change from baseline, immediately after completion of study treatment, and 100 days post-transplant
  Perceived Social Support from Friends (PSS-Fr) is a self-report scale using 3-point rating responses ranging from 0 to 2 designed to measure the extent to which individuals perceive that their needs for support, information, and feedback are fulfilled by friends.
Assess changes in perceived social support from family | Change from baseline, immediately after completion of study treatment, and 100 days post-transplant
  Perceived Social Support from Family (PSS-Fa) is a self-report, 3-point response (Yes, No, I don't know) scale, designed to measure the extent to which individuals perceive that their needs for support, information and feedback are fulfilled by family.
Assess changes in perceived social support from healthcare providers | Change from baseline, immediately after completion of study treatment, and 100 days post-transplant
  Perceived Social Support from Health Care Providers (PSS-HCP) is a self-report, 3-point rating scale adapted by Haase from items on the Perceived Social Support-Friends scales102 to correspond to health care provider relationships. Items indicate the extent to which individuals perceive their needs for support, information, and feedback are fulfilled by health care providers.
Assess changes in Hope from stem cell transplantation (STC) experience: | Change from immediately after completion of study treatment, and 100 days post-transplant
  Measured by indicators of hope. Herth Hope Index (HHI) items are on a 4-point scale, ranging from 1 (strongly disagree) to 4 (strongly agree); higher summative scores indicate greater hope.
Assess changes in Spiritual Perspective from stem cell transplantation (STC) experience | Change from immediately after completion of study treatment, and 100 days post-transplant
  Measured by indicators spiritual perspective. Reed Spiritual Perspective Scale (RSPS) is a one-factor scale that measures the saliency of spiritual beliefs and behaviors in the respondent's life.157 The response format is a 6-point Likert scale anchored with words describing the frequency of behaviors.
Assess changes of Higher Resilience: Haase Adolescent Resilience in Cancer Scale | Change from after completion of study treatment and 100 days post-transplant
  Haase Adolescent Resilience in Cancer Scale measures resilience related to illness. The scale uses a 6-point Likert-type scale ranging form: 1 (strongly disagree) to 4 (strongly agree); higher summative scores indicate greater resilience. Validity of the scales was found in predictive correlations with self-esteem, self-transcendence, confidence/mastery and quality of life. In Haase's preliminary studies, alpha reliability coefficients were 0.84 - 0.86.
Assess changes of Higher Resilience (self esteem, confidence, self-transcendence): NCS | Change from after completion of study treatment, and 100 days post-transplant
  Nowotny Confidence Subscale (NCS) of the Nowotny Hope Scale is a self-report of confidence in one's own ability, which uses a 4-point Likert response format of strongly agree to strongly disagree
Assess changes of Higher Resilience (self esteem, confidence, self-transcendence): STS | Change from after completion of study treatment, and 100 days post-transplant
  Reed Self-Transcendence Scale (STS) assesses activities and perspectives individuals engage in to expand their boundaries via 4-point Likert response scales
Assess changes in Higher Resilience (self esteem, confidence, self-transcendence): SES | Change from after completion of study treatment, and 100 days post-transplant
  Rosenberg Self-esteem Scale (SES) measures attitudes toward one's self. Responses are on a 4-point Likert scale.
Assess changes in indicators of well-being and global quality of life: LASA Uniscale | Change from baseline, immediately after completion of study treatment, and 100 days post-transplant
  Measured by indicators of well-being and global quality of life.LASA Uniscale is a global QOL self-report one-item instrument: "Please score how you feel your life has been affected by the state of your health (any disease or treatment) during the last week".160 The item is adopted from the Southwest Oncology Group protocol, which adapted the scale from a linear analogue to categorical format with 5 response categories ranging from extremely unpleasant to normal (no change).
Assess changes in indicators of well-being and global quality of life: IWB | Change from baseline, immediately after completion of study treatment, and 100 days post-transplant
  Measured by indicators of well-being and global quality of life. Index of Well-being (IWB) is a semantic differential scale describing present life using adjective extremes such as discouraging/hopeful.

SECONDARY OUTCOMES:
Qualitatively describe the perception of helpfulness and meaningfulness of both the low-dose and TMV interventions for AYA and family members | 100 days post-transplant
  The Interview Guide is used to collect data to answer research questions. The interview schedule includes open-ended questions. Examples of questions for the TMV group AYA and designated caregiver, respectively, are: "Tell me about your experience of being involved in the music video production" and "Tell me what you think it meant for your adolescent to complete the video." (Appendix 1) The interview proceeds until the participant feels the experience is fully described

CONTACTS AND LOCATIONS:
Overall Officials: Joan E Haase, Principal Investigator — Children's Oncology Group
Locations (3):
- United States (3):
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Children's Oncology Group, Philadelphia, Pennsylvania